CLINICAL TRIAL: NCT05002764
Title: Differential Vulnerability of Individual Thalamic Nuclei: Toward New Biomarkers in Multiple Sclerosis
Brief Title: Thalamic Nuclei Volumes in Multiple Sclerosis
Acronym: THALNUC-MS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/33
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Thalamus; Nuclei; Atrophy
MeSH Terms: conditions — Multiple Sclerosis; Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The thalamus is composed of several nuclei interlocked in a complex anatomy. In multiple sclerosis (MS), the thalamus can be altered due to disconnection by white matter lesions and due to direct damages that could be partly mediated by CSF. Due to such pathophysiology and complex anatomy, some nuclei could be more vulnerable to multiple sclerosis than others. We will test this hypothesis by using a new algorithm to automatically segment several nuclei that we will be applied to the French national MS database

ELIGIBILITY:
Inclusion Criteria :

* Patient older than 18 years old.
* With Multiple Sclerosis according to Mc Donald 2017 criteria or with clinically isolated syndrome and included with OFSEP cohort.
* Phenotype known (RR, SP, PP or CIS).
* Date of diagnosis known.
* With at least one MRI that includes 3D T1 and FLAIR at 1.5T or 3T.

Exclusion Criteria :

* Stroke
* Other causes of dementia not caused by Multiple Sclerosis (Alzheimer's disease, Parkinsonian syndromes…)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Sclerosis and at least one MRI that includes 3D T1 and FLAIR at 1.5T or 3T.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Volume of thalamic nuclei | At inclusion in the cohort
  Volume of individual thalamic nuclei according to disease duration.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France